CLINICAL TRIAL: NCT01069107
Title: Acute Admission to Hallingdal Sjukestugu. Can Acute Admissions to a Community Hospital be a Realistic Alternative to General Hospital Admissions?
Brief Title: Acute Admission to Hallingdal Sjukestugu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Sor-Ost (Other Government)
Collaborators: Ringerike sykehus, Vestre Viken HF (Unknown); University of Oslo (Other); Norwegian University of Science and Technology (Other)
Responsible Party: Principal Investigator, Oystein Lappegard, Forsker, Helse Sor-Ost
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 09-1300 REK; 20100101 (Other: Helse Sorost)
Record Dates: First submitted 2010-02-04; First posted 2010-02-17 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Morbidity; Health Economy; Quality
Keywords: community hospital; alternative acute admissions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Consume of health services (Active Comparator): One year follow-up of patients randomized to two different levels of health care
  Interventions: Other: Cottage Hospital Care

INTERVENTIONS:
Other: Cottage Hospital Care — Care at a cottage hospital compared with care at a general hospital

SUMMARY:
The main objective of the project is to assess whether a community hospital may have or should have a role in the Norwegian health care system in the acute treatment of a defined group of patients.

DETAILED DESCRIPTION:
The research project's objective is to analyze whether acute admissions to Hallingdal sjukestugu (HSS) is a real alternative to hospitalization in a general hospital.

HSS is a community hospital and a department under Ringerike General Hospital (RS) and is located in Hallingdal 170 km from the RS. It is an established practice that the general practitioners in Hallingdal send selected patients in need for acute treatment to HSS in place of RS. In 2008 this accounted for 10.1% of the total number of acute inpatients from the six municipalities of Hallingdal.

The research program includes a prospective, randomized study in which all patients intended for acute inpatient at HSS are distributed randomly into two groups, an intervention group who is admitted to HSS, and a control group who is sent to RS. A minimum of 70 patients are included in each group.

The patients are going to be followed through one year after the hospital stay and all contacts with the specialist health services and the municipal health care services will be registered. There will also be collected data on the patients' functioning level and the patients' opinion about quality of the hospital stay. Through standardized questionnaire the involved health professional will be asked about their reviews.

Three studies will analyze the patients' progress, economics and quality in the two groups. The three studies will together constitute a doctoral thesis.

The research project will provide a better basis for assessing the role of local medical centers in the Norwegian health care in the acute treatment of a defined group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who by the general practitioner are intended for acute admission to HSS and where the specialist on call at RS approves such admissions.
* Patients residing in Hallingdal municipalities.

Exclusion Criteria:

* Patients with injuries and acute and/or unclear illnesses in need of diagnosis, treatment or monitoring in an acute hospital.
* Urgent births at HSS.
* Acute psychiatric admissions to hospital.
* Patients with serious mental disorders.
* Patients who during the follow-up year move to a municipality outside of Hallingdal.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2010-04; Primary Completion 2013-04 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
A triangulation of patient health consequences, patients' perceived quality and a health economy analyses. | One year

SECONDARY OUTCOMES:
All contacts with the specialist health services and the municipal health care services will be registered. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Per Hjortdahl, Prof., Study Director — Institute of General Practice and Community Medicine , University of Oslo
Locations (1):
- Hallingdal sjukestugu, Ål, Buskerud, Norway

REFERENCES:
- [Derived] Lappegard O, Hjortdahl P. Acute admissions to a community hospital - health consequences: a randomized controlled trial in Hallingdal, Norway. BMC Fam Pract. 2014 Dec 10;15:198. doi: 10.1186/s12875-014-0198-1. PMID 25491726